CLINICAL TRIAL: NCT06401538
Title: An Open-Label Phase 2 Study to Evaluate the Efficacy, Safety and Tolerability of BMB-101 in Adults With Either Classic Absence Epilepsy (With or Without Eyelid Myoclonia (EEM; Jeavons Syndrome), OR Developmental Epileptic Encephalopathy (DEE).
Brief Title: BMB-101 in Absence Epilepsy and DEE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bright Minds Biosciences Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMB-101-103
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Absence Epilepsy; Jeavons Syndrome; Dravet Syndrome; Lennox Gastaut Syndrome
MeSH Terms: conditions — Epilepsy, Absence; Epilepsies, Myoclonic; Lennox Gastaut Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMB-101 (Experimental): BMB-101 10 mg/ml liquid
  Interventions: Drug: BMB-101

INTERVENTIONS:
Drug: BMB-101 — BMB-101 liquid administered orally twice a day for 3 months

SUMMARY:
The study is a pilot, open-label, study to test whether BMB-101 is safe and effective in reducing the frequency of seizures in subjects with Absence Epilepsy including Epilepsy with Eyelid Myoclonia (also called Jeavons Syndrome) as well as Developmental Epileptic Encephalopathies such as Dravet and Lennox Gastaut. The study will last up to 6 months. There will be a 1 month screening period, then up to 3 months on open-label BMB-101 including titration and tapering/washout periods, and then a 1 month follow-up period. There will be 6 clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a diagnosis of Absence Epilepsy with or without eyelid myoclonia (Jeavons Syndrome) or a diagnosis of Developmental and Epileptic Encephalopathy (DEE) such as Dravet syndrome or Lennox-Gastaut syndrome or other DEE.
2. Subjects with Absence must experience at least 4 episodes of 3-4/second SWD lasting at least 3 seconds each in a 24 hour EEG during the baseline period. Those with DEE must have a typical EEG pattern for DEE on routine EEG and experience at least 4 seizures during the 4 week baseline period prior to BMB-101 administration.
3. Subjects can be male or female ages 18-65 inclusive at time of baseline.
4. Subject must have tried at least one anti-seizure medication at a recommended dose and duration and must be on a stable dose on their current anti-seizure medications for at least 4 weeks prior to baseline and remain stable throughout the study.
5. Subjectis willing and able to be compliant with diary completion, visit schedule, and study drug accountability.
6. Female subjects of childbearing potential must have a negative urine pregnancy test at baseline. Subjects of childbearing or child-fathering potential must be willing to use medically acceptable forms of birth control, which includes abstinence, while in this study and for 90 days after the last dose of study drug.

Exclusion Criteria:

1. Subject has current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, pulmonary hypertension, myocardial infarction or stroke, or clinically significant structural cardiac abnormality.
2. Subject has moderate or severe hepatic impairment. Asymptomatic subjects with mild hepatic impairment (elevated liver enzymes < 3x upper limit of normal (ULN) and/or elevated bilirubin <2x ULN) may be entered into the study after review and approval by the Medical Monitor in conjunction with the sponsor, in consideration of comorbidities and concomitant medications.
3. Subject has severe renal impairment (estimated glomerular filtration rate <30mL/min/1.73m2)
4. Clinically significant ECG abnormality such as QTcF >450 msec (males) or >470 msec (females)
5. Subject is receiving concomitant therapy with: fenfluramine, lorcaserin, monoamine-oxidase inhibitors, SSRIs, SNRIs, tricyclic antidepressants or other serotonergic agonists or antagonists (antipsychotics).
6. Subject is currently receiving an investigational medicinal product.
7. Subject has participated in another clinical trial within the past 30 days (calculated from that study's last scheduled visit). Participation in non-treatment trials will be reviewed by the medical monitor.
8. Subject has a history of drug or alcohol abuse within the last 12 months or a positive urine drug screen (with the exception of cannabinoids).
9. A current C-SSRS score of 4 or 5 at baseline or history of suicide attempt at any time during the past year
10. Subject has a clinically significant condition or has had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to the Baseline Visit, other than epilepsy, that would negatively impact study participation, collection of study data, or pose a risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in seizure frequency in DEE subjects | 10 weeks
  Seizure diary
Change from baseline in the number of generalized spike-wave discharges (GSWD) on the 24 hr EEG in Absence subjects. | 6 weeks
  24 hour EEG

SECONDARY OUTCOMES:
Change from baseline in quality of life | 6-10 weeks
  Quality of Life in Epilepsy (QOLIE-31) for adults

CONTACTS AND LOCATIONS:
Overall Officials: Terence O'Brien, MD, Principal Investigator — The Alfred
Locations (5):
- Australia (5):
  - The Prince of Wales Hospital, Randwick, New South Wales
  - Royal Brisbane and Womans Hospital, Herston, Queensland
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No